CLINICAL TRIAL: NCT03339076
Title: A Prospective Evaluation of the Catheter Science M3 "Mini Catheter" for Patients With Prostatic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Gaines W. Hammond Jr. MD FACS (Individual)
Responsible Party: Sponsor-Investigator, Dr. Gaines W. Hammond Jr. MD FACS, INVESTIGATOR - SPONSOR, Hammond, Gaines W., Jr., M.D. FACS
Organization: Hammond, Gaines W., Jr., M.D. FACS (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study # 17/10/04
Record Dates: First submitted 2017-10-24; First posted 2017-11-13 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-11

CONDITIONS: Urinary Retention
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Intervention Model Description: This single arm prospective study is designed to produce valid scientific evidence regarding safety and efficacy of the M3 in establishing urinary drainage and allowing the control of micturition when indwelling for <28 days in male patients. The total study population will initially include 50 subjects with open enrollment of additional subjects.
  1. Study Timeline and Calendar
  The maximum indwelling time for the DEVICE should be <28 days, at which time the DEVICE will be removed, and the patient will be offered the option of insertion of a new M3 Catheter or return to the bladder drainage technique used prior to M3 Catheter insertion. All patients will be followed until patient is off study or until end of study, whichever occurs first.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- For a single-arm trial (Other): Inclusion Criteria with intervention replacing either a foley catheter or self intermittent catheter with the M3 "Mini Catheter"
  1. Males > 50 years of age
  2. Signed subject informed consent
  3. Patients with actual urinary retention dependent on Foley Catheter or Intermittent Catheter
  4. Inclusion will start once the M3 is placed and a functioning bladder is demonstrated.
  Exclusion Criteria
  1. Inability to undergo bladder catheterization with the M3 due to anatomical challenges (i.e. urethral stricture, bladder neck contracture, false passage or false passages or other history of urethral stricture)
  2. Gross hematuria
  3. Hypotonic Neurogenic Bladder (the placement of the M3 may isolate the cause of the retention with the bridging of the prostate as bladder dysfunction rather than prostate obstruction).
  Interventions: Device: M3 "MINI CATHETER"

INTERVENTIONS:
Device: M3 "MINI CATHETER" — Participants in the study are using either a foley catheter or Clean Intermittent Catheter devices to facilitate bladder drainage. The study is an alternative method of facilitating bladder drainage with the M3 "Mini Catheter."

SUMMARY:
The Catheter Science M3 "Mini Catheter" has been developed for management of urinary retention. This temporary device allows for normal functioning of the external striated sphincter. The design contributes to its atraumatic insertion and removal. It is a short catheter segment which is attached to a monofilament suture which runs thru the lumen of the urethra and is attached to a small plastic "bobber". This study is designed to validate the reduction in these adverse effects: The suture to the outside allows for repositioning should the device slip back into the bladder and facilitates removal. With volitional voiding and competent external sphincter, patients are able to void spontaneously without the need of a collection device and are continent. The design enhances the flow characteristics and reduces post void residual. Since the M3 does not have a tubular segment thru the tip of the penis or sphincter, biofilm production is eliminated.

DETAILED DESCRIPTION:
This single arm, prospective study is designed to produce valid scientific evidence regarding:

1. Safety and efficacy of the Catheter Science M3 "Mini Catheter" in establishing urinary drainage and allowing the control of micturition when indwelling for a period of time up to but less than 28 days in male patients with prostate outlet obstruction who have been dependent on either a Foley catheter or Intermittent Catheterization.
2. The study purpose is to measure the rate of catheter-related urinary tract infections in patients with the M3 in place as compared to the known infection rate for patients with a Foley catheter in place over the same period of time.

A single arm study design was chosen because there is no alternative treatment to serve as an appropriate control. The M3 de-obstructs the prostatic urethra, allows volitional voiding function in patients with a contractile bladder. A Foley catheter, a pre- amendment device, was considered for a control treatment. Although a Foley catheter is used to establish urinary drainage initially with close to 100% efficacy, it does not allow for voluntary micturition as defined with the coordination of contraction of the bladder with the relaxation of the striated external sphincter. The ability of the bladder to fill and contract with a Foley is altered. The M3 allows for the bladder to fill since the sphincter is not bridged. Volitional micturition is initiated with bladder contraction coordinated with a relaxation of the external striated sphincter. The flow of urine is thru and around the M3 rather than only intraluminal in the Foley. The direction of urine flow with the M3 is in one direction in contrast to the Foley catheter and external collection device which is bi-directionally. The flow of urine back into the bladder has long been viewed as a significant contributor to the CAUTI. The Foley is a passive drainage device which simply drains the bladder with negative pressure produced in a closed system aided with gravity. The laterally placed intake eyes of the Foley are vulnerable to occlusion of the bladder mucosa being pulled into the lumen by the negative pressure of the closed system. The requirement of an external collecting bag coupled with the Foley traversing the entire length of the Urethra, severely impairs activities of daily life. The comparative lifestyle changes between the Foley Catheter, Intermittent Catheter and M3 group is not the focus of this study of the Safety and Efficacy characteristics of the M3 vs Foley comparison, but will be obvious to patients and clinicians.

The retention balloon inflation channel impacts the internal diameter of the Foley. The Balloon prevents complete emptying of the bladder with resultant residual of 10-100cc reported. Since there is no consistent flow of urine around a Foley to help "wash out bacteria" the formation of biofilm is accelerated. The Foley violates the anatomical protective points (penile meatus, sphincter, prostatic urethral and bladder neck) which help prevent bacterial contamination. The M3 CAUTI reduction as compared to the Foley and Intermittent Catheter Group is due to a series of important design features. The removal of a retention balloon allows for the internal diameter to be enlarged. The 3 wings Malecott promotes retention of the device as well as preventing bladder mucosal plugging of the lumen during voiding contractions. This design also promotes an improved post void residual compared to a Foley device. The residual urine in the bladder with a Foley as well a slow flow rate promotes encrustations and occlusion of the Foley.

ELIGIBILITY:
Inclusion Criteria:

* Males > 50 years of age
* Signed subject informed consent (see Appendix "A")
* Patients with actual urinary retention dependent on Foley Catheter or Intermittent Catheter
* Inclusion will start once the M3 is placed and a functioning bladder is demonstrated.

Exclusion Criteria:

* Inability to undergo bladder catheterization with the M3 due to anatomical challenges (i.e. urethral stricture, bladder neck contracture, false passage or false passages or other history of urethral stricture)
* Gross hematuria
* Hypotonic Neurogenic Bladder (the placement of the M3 may isolate the cause of the retention with the bridging of the prostate as bladder dysfunction rather than prostate obstruction).

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The percentage of Catheter Acquired Urinary Tract Infections with the M3 Mini Catheter. | Time of placement up to 28 days.
  1.The study purpose is to measure the rate of catheter-related urinary tract infections in patients with the M3 in place as compared to the known infection rate for patients with a Foley catheter in place over the same period of time.
The percentage of M3 removed due to encrustation and blockage of the M3. | Weekly from time of placement up to 28 days.
  The percentage of M3 devices removed due to urinary retention caused by device encrustation.
Measurement of Bladder Drainage | Weekly from time of placement up to 28 days.
  The Post Void Residual after M3 placement
Flow Rate after M3 placement | At time of placement and weekly up to 28 days.
  The flow rate after M3 placement with a bladder volume of at least 120 cc.

SECONDARY OUTCOMES:
Failure of the M3 as a choice of bladder drainage over Foley Catheter or Self Intermittent Catheter drainage | From time of Placement up to 28 days.
  The failure of the M3 to drain the bladder with the requirement to reinstitute Foley Drainage or Self Intermittent Catheter by choice versus M3 Mini Catheter

CONTACTS AND LOCATIONS:
Overall Officials: GAINES W HAMMOND, MD, Principal Investigator — Watson Clinic Center for Research, Inc.
Locations (1):
- Watson Clinic Llp, Lakeland, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After completion of the study anticipated to be in March 2018 for a 2 year period of time.
Access Criteria: Appropriate credentials to access material with the identifying markers of patients identity withheld.